CLINICAL TRIAL: NCT02368366
Title: Comparative Effectiveness of Family Problem-Solving Therapy (F-PST) for Adolescent TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Case Western Reserve University (Other); Children's Hospital Colorado (Other); MetroHealth Medical Center (Other); Nationwide Children's Hospital (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-1306-02435
Record Dates: First submitted 2014-10-27; First posted 2015-02-23 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Tbi; Intracranial Edema; Brain Edema; Craniocerebral Trauma; Head Injury; Brain Hemorrhage, Traumatic; Subdural Hematoma; Brain Concussion; Head Injuries, Closed; Epidural Hematoma; Cortical Contusion; Wounds and Injuries; Disorders of Environmental Origin; Trauma, Nervous System; Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Craniocerebral Trauma; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Brain Concussion; Head Injuries, Closed; Hematoma, Epidural, Spinal; Brain Contusion; Wounds and Injuries; Disorders of Environmental Origin; Trauma, Nervous System; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Therapist Guided Face to Face FPST (Experimental): Therapist Guided Face to Face Family Problem Solving Families assigned to this arm will meet with the therapist in person at the medical center TBI clinic. Sessions will last approximately 60 minutes and cover didactic content using printed handouts provided as part of a family workbook.
  Interventions: Behavioral: Therapist Guided Face to Face Family Problem Solving
- Therapist Guided Online FPST (Experimental): Therapist Guided Online Family Problem Solving Families assigned to this arm will receive a password enabling them to access the online intervention materials throughout the course of the intervention. Each session of online F-PST consists of a self-guided online portion providing didactic content regarding the desired skill (i.e., problem-solving), video clips showing individuals and families modeling the skill, and exercises and assignments giving the family an opportunity to practice the skill. During synchronous, videoconference sessions with the therapist, the family will review the online materials and practice the problem-solving process.
  Interventions: Behavioral: Therapist Guided Online Family Problem Solving
- Self-Guided Online FPST (Experimental): Self-Guided Online Family Problem Solving Families in the self-guided, online F-PST arm will receive a password enabling them to access the online intervention materials throughout the course of the intervention. They will receive access to the same web-modules as the therapist-guided group, but will review them on their own without therapist support. Participants in this group will be encouraged to complete web modules at the same schedule as participants in the other groups. If the family fails to log on or complete web modules, they will receive reminders via phone, text, or e-mail.
  Interventions: Behavioral: Self-Guided Online Family Problem Solving

INTERVENTIONS:
Behavioral: Therapist Guided Face to Face Family Problem Solving — Families assigned to this arm will meet with the therapist in person at the medical center TBI clinic. Sessions will last approximately 60 minutes and cover didactic content using printed handouts provided as part of a family workbook.
  Arms: Therapist Guided Face to Face FPST
Behavioral: Therapist Guided Online Family Problem Solving — Families assigned to this arm will receive a password enabling them to access the online intervention materials throughout the course of the intervention. Each session of online F-PST consists of a self-guided online portion providing didactic content regarding the desired skill (i.e., problem-solving), video clips showing individuals and families modeling the skill, and exercises and assignments giving the family an opportunity to practice the skill. During synchronous, videoconference sessions with the therapist, the family will review the online materials and practice the problem-solving process.
  Arms: Therapist Guided Online FPST
Behavioral: Self-Guided Online Family Problem Solving — Families in the self-guided, online F-PST arm will receive a password enabling them to access the online intervention materials throughout the course of the intervention. They will receive access to the same web-modules as the therapist-guided group, but will review them on their own without therapist support. Participants in this group will be encouraged to complete web modules at the same schedule as participants in the other groups. If the family fails to log on or complete web modules, they will receive reminders via phone, text, or e-mail.
  Arms: Self-Guided Online FPST

SUMMARY:
Traumatic brain injury (TBI) is the most common cause of acquired disability in youth and a source of significant morbidity and family burden. Novel behavior problems are among the most common and problematic consequences, yet many youth fail to receive needed psychological services due to lack of identification and access. Linking youth with TBI to effective treatments could improve functional outcomes, reduce family burden, and increase treatment satisfaction. The investigators overarching aim is to compare the effectiveness, feasibility, and acceptability of three formats of family problem solving therapy (F-PST) for improving functional outcomes of complicated mild to severe adolescent TBI: therapist-guided, face-to-face; therapist-guided online; and self-guided, online F-PST.

DETAILED DESCRIPTION:
Background: Traumatic brain injury (TBI) is the most common cause of acquired disability in youth and a source of significant morbidity and family burden. Novel behavior problems are among the most common and problematic consequences, yet many youth fail to receive needed psychological services due to lack of identification and access. Linking youth with TBI to effective treatments could improve functional outcomes, reduce family burden, and increase treatment satisfaction.

Methods: The investigators overarching aim is to compare the effectiveness, feasibility, and acceptability of three formats of family problem solving therapy (F-PST) for improving functional outcomes of complicated mild to severe adolescent TBI: therapist-guided, face-to-face; therapist-guided online; and self-guided, online F-PST. The efficacy of face-to-face and online F-PST in reducing behavior problems following TBI has been established. However, their comparative acceptability and effectiveness are unknown and it is unclear if families could also benefit from online F-PST without therapist support. To identify which patients benefit most from each intervention, participants will be stratified by distance from the clinic with patients living more than 20 miles or 60 minutes from the clinic randomized to one of the two online arms and others equally randomized among three arms. Patient-reported outcomes pertaining to child, caregiver, and family functioning along with patient treatment preferences will be assessed: prior to treatment initiation, at treatment completion, and at a follow-up 3 months later. Stakeholder input (adolescents with TBI and their caregivers) will guide measurement selection and refinements to the treatment protocols. Each treatment modality consists of 10-14 sessions addressing TBI education, problem-solving, self-regulation, and family communication, but varies in the nature and extent of therapist involvement. Participants will include families of 120 adolescents age 14-18 recruited from four metropolitan TBI centers. Mixed models analyses will be used to examine group differences in improvements in child behavior/functioning, caregiver distress, and family burden. Moderators of comparative effectiveness including socioeconomic status, prior technology use, and patient preferences will be examined.

Anticipated Impact: Results will elucidate the relative effectiveness of face-to-face versus online and self-directed versus therapist-supported online modes of treatment including patient and family preferences. They will also provide information about how these programs can be delivered and disseminated through existing head injury follow-up clinics. These data could potentially be translated to other patient populations of youth with psychological symptoms arising from neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe TBI
* Overnight hospital stay
* English-speaking
* Parent must be willing to provide informed consent

Exclusion Criteria:

* Child does not live with parents or guardian
* Child or parent has history of hospitalization for psychiatric problem
* Child suffered a non-blunt injury (e.g., projectile wound, stroke, drowning, or other form of asphyxiation)
* Diagnosed with moderate or severe mental retardation, autism, or a significant developmental disability

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, post-intervention and 3 months post-intervention

SECONDARY OUTCOMES:
Center for Epidemiology Scale for Depression (CES-D) | Baseline, post-intervention and 3 months post-intervention
Health and Behavior Inventory (HBI) | Baseline, post-intervention and 3 months post-intervention
Ohio State University (OSU) Traumatic Brain Injury (TBI) Identification Method (OSU TBI-ID) | Baseline
Brief Symptom Inventory (BSI) | Baseline, post-intervention and 3 months post-intervention
Strengths and Difficulties Questionnaire (SDQ) | Baseline, post-intervention and 3 months post-intervention
Pediatric Quality of Life Inventory (PedsQL) | Baseline, post-intervention and 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shari Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - The Children's Hospital, Denver, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Wade SL, Cassedy AE, Taylor HG, McNally KA, Kirkwood MW, Stancin T, Horn PS, Kurowski BG. Adolescent quality of life following family problem-solving treatment for brain injury. J Consult Clin Psychol. 2019 Nov;87(11):1043-1055. doi: 10.1037/ccp0000440. Epub 2019 Sep 26. PMID 31556652